CLINICAL TRIAL: NCT02048917
Title: Optimization of Smoking Cessation Strategies Concurrent With Treatment of Tobacco Related Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Kentucky (Other)
Collaborators: Kentucky Lung Cancer Research Program (Other)
Responsible Party: Principal Investigator, Joseph Valentino, Study Chair, University of Kentucky
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-13-MULTI-13-KCTN-1301; KCTN-1301 (Other: Markey Cancer Center)
Record Dates: First submitted 2014-01-27; First posted 2014-01-29 (Estimated); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Lung Cancer; Head and Neck Cancer
Keywords: Smoking; Cessation; Bupropion; Varenicline; Nicotine; Counseling; Tobacco
MeSH Terms: conditions — Lung Neoplasms; Head and Neck Neoplasms; Smoking | interventions — Bupropion; Varenicline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- High Intensity Counseling + Long Acting NRT + PRN NRT (Experimental): High Intensity Counseling + Long Acting NRT + PRN NRT
  Interventions: Drug: High Intensity Counseling + Long Acting NRT + PRN NRT
- High Intensity Counseling + bupropion + PRN NRT (Experimental): High Intensity Counseling + bupropion + PRN NRT
  Interventions: Drug: High Intensity Counseling + bupropion + PRN NRT
- High Intensity Counseling + varenicline + PRN NRT (Experimental): High Intensity Counseling + varenicline + PRN NRT
  Interventions: Drug: High Intensity Counseling + varenicline + PRN NRT
- High Intensity Counseling + Long Acting NRT (Experimental): High Intensity Counseling + Long Acting NRT
  Interventions: Drug: High Intensity Counseling + Long Acting NRT
- High Intensity Counseling + bupropion (Experimental): High Intensity Counseling + bupropion
  Interventions: Drug: High Intensity Counseling + bupropion
- High Intensity Counseling + varenicline (Experimental): High Intensity Counseling + varenicline
  Interventions: Drug: High Intensity Counseling + varenicline
- Low Intensity Counseling + Long Acting NRT + PRN NRT (Experimental): Low Intensity Counseling + Long Acting NRT + PRN NRT
  Interventions: Drug: Low Intensity Counseling + Long Acting NRT + PRN NRT
- Low Intensity Counseling + bupropion + PRN NRT (Experimental): Low Intensity Counseling + bupropion + PRN NRT
  Interventions: Drug: Low Intensity Counseling + bupropion + PRN NRT
- Low Intensity Counseling + varenicline + PRN NRT (Experimental): Low Intensity Counseling + varenicline + PRN NRT
  Interventions: Drug: Low Intensity Counseling + varenicline + PRN NRT
- Low Intensity Counseling + Long Acting NRT (Experimental): Low Intensity Counseling + Long Acting NRT
  Interventions: Drug: Low Intensity Counseling + Long Acting NRT
- Low Intensity Counseling + bupropion (Experimental): Low Intensity Counseling + bupropion
  Interventions: Drug: Low Intensity Counseling + bupropion
- Low Intensity Counseling + varenicline (Experimental): Low Intensity Counseling + varenicline
  Interventions: Drug: Low Intensity Counseling + varenicline

INTERVENTIONS:
Drug: High Intensity Counseling + Long Acting NRT + PRN NRT — High Intensity Counseling + Long Acting NRT + PRN NRT
  Arms: High Intensity Counseling + Long Acting NRT + PRN NRT
Drug: High Intensity Counseling + bupropion + PRN NRT — High Intensity Counseling + bupropion + PRN NRT
  Arms: High Intensity Counseling + bupropion + PRN NRT
Drug: High Intensity Counseling + varenicline + PRN NRT — High Intensity Counseling + varenicline + PRN NRT
  Arms: High Intensity Counseling + varenicline + PRN NRT
Drug: High Intensity Counseling + Long Acting NRT — High Intensity Counseling + Long Acting NRT
  Arms: High Intensity Counseling + Long Acting NRT
Drug: High Intensity Counseling + bupropion — High Intensity Counseling + bupropion
  Arms: High Intensity Counseling + bupropion
Drug: High Intensity Counseling + varenicline — High Intensity Counseling + varenicline
  Arms: High Intensity Counseling + varenicline
Drug: Low Intensity Counseling + Long Acting NRT + PRN NRT — Low Intensity Counseling + Long Acting NRT + PRN NRT
  Arms: Low Intensity Counseling + Long Acting NRT + PRN NRT
Drug: Low Intensity Counseling + bupropion + PRN NRT — Low Intensity Counseling + bupropion + PRN NRT
  Arms: Low Intensity Counseling + bupropion + PRN NRT
Drug: Low Intensity Counseling + varenicline + PRN NRT — Low Intensity Counseling + varenicline + PRN NRT
  Arms: Low Intensity Counseling + varenicline + PRN NRT
Drug: Low Intensity Counseling + Long Acting NRT — Low Intensity Counseling + Long Acting NRT
  Arms: Low Intensity Counseling + Long Acting NRT
Drug: Low Intensity Counseling + bupropion — Low Intensity Counseling + bupropion
  Arms: Low Intensity Counseling + bupropion
Drug: Low Intensity Counseling + varenicline — Low Intensity Counseling + varenicline
  Arms: Low Intensity Counseling + varenicline

SUMMARY:
The purpose of this study is to find an optimal smoking cessation strategy in patients undergoing therapy for lung and head and neck cancers at selected cancer centers in Kentucky by delivering high quality smoking cessation to all enrolled patients. This study will also examine the feasibility of routinely implementing an array of smoking cessation strategies for this patient population.

DETAILED DESCRIPTION:
Subjects enrolled in the study will be placed in one of twelve treatment arms. Subjects in each of the twelve treatment regimens will receive either varenicline or bupropion or long-acting nicotine replacement therapy, with or without use of supplemental nicotine replacement therapy, and in combination with either standard of care smoking cessation counseling or high intensity/motivational smoking cessation counseling.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥ 18 years of age.
* Patient with newly diagnosed or recurrent, histologic diagnosis of any of the following tobacco related malignancies:

  1. Lung or Bronchus cancer or Head & Neck, cancers (all sites).
  2. Esophagus, Stomach, Pancreas, Kidney, Urinary Bladder, Colon, Rectum, Cervix, Vulvar, Vaginal
  3. Carcinoma in situ undergoing definitive surgical resection or treatment (ex: radiation of the larynx, and gynecologic tract hysterectomy, vulvectomy - except gynecologic patients undergoing ablative or local excisional therapies [laser ablation,cervical conization, LEEP].
* Having smoked at least 1 cigarette within 4 weeks of study enrollment.
* Having at least a 10-pack year history of cigarette smoking.
* Having smoked at least one cigarette within 1 month of cancer diagnosis.
* Life expectancy is greater than 1 year.
* Patient has an AUDIT score of < 10.
* Patient has ECOG Performance Status of <=2.
* Patients must have the ability to understand and the willingness to provide signed written informed consent document.

Exclusion Criteria:

* Known allergy attributed to bupropion, varenicline, transdermal or lozenge nicotine.
* History of suicide attempt or preparation for attempt within the past 10 years.
* C-SRSS Baseline/Screening:

  1. Patient response of "Yes" to any question except question 1.
  2. Patient response of "Yes" to any question in column one (lifetime), except question 1, is not exclusionary unless judged by the investigator to be significant in ideation, intensity, behavior or attempts, and precludes participation.
* Hospitalized for psychiatric illness within the past two years.
* History of Bipolar disorder.
* Currently taking Bupropion for depression.
* Patient has taken monoamine oxidase inhibitors (MAOI) in the past two weeks.
* History of eating disorder such as anorexia or bulimia.
* Active widespread skin disorders such as psoriasis, chronic urticarial or dermatitis
* History of epilepsy or seizure disorder.
* Active severe kidney or liver disease.
* Women must not be pregnant or lactating. Women of reproductive-potential must have negative serum or urine pregnancy test within 7 days prior to study enrollment and agree to use method of contraception during and for 30 days following last cessation drug dose.
* Patients within three months of a myocardial infarction.
* Patients with unstable angina or serious arrhythmia.
* Patients with psychiatric disability judged by the investigator to be clinically significant so as to preclude informed consent or compliance with drug intake.
* Patient taking varenicline or bupropion within one month of study enrollment.
* Participation in any other investigational drug study within 4 weeks of study enrollment.
* Currently enrolled in other professional tobacco cessation therapeutic intervention.
* Enrollment in a concurrent cancer therapeutic trial will require prior review and approval by the study site PI to determine that there are no drug interactions concerns.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2014-07-22 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
Cigarette use | 8 weeks
  Seven day point prevalence of cigarette use confirmed with CO testing at eight weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Valentino, M.D., Principal Investigator — University of Kentucky
Locations (10):
- United States (10):
  - King's Daughters Medical Center, Ashland, Kentucky
  - Hardin Memorial Health Cancer Care Center, Elizabethtown, Kentucky
  - ARH Cancer Center, Hazard, Kentucky
  - Kentucky Cancer Clinic, Hazard, Kentucky
  - Lexington Veterans Affair Medical Center, Lexington, Kentucky
  - University Of Kentucky, Markey Cancer Center, Lexington, Kentucky
  - University of Louisville, James Graham Brown Cancer Center, Louisville, Kentucky
  - St. Claire Regional Medical Center, Morehead, Kentucky
  - Owensboro Health, Owensboro, Kentucky
  - St. Mary's Medical Center, Huntington, West Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273